CLINICAL TRIAL: NCT06797492
Title: Virtual Reality for Shoulder Rehabilitation: New Approaches and Applications in Orthopedics
Brief Title: Virtual Reality for Shoulder Rehabilitation
Acronym: REVISA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Umile Giuseppe Longo, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 234.24 CET2 cbm; PNC0000007 - CUP: B53C22006980 (Other Grant/Funding Number: Italian Ministry of Research, under the complementary actions to the NRRP "Fit4MedRob - Fit for Medical Robotics")
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Musculoskeletal Disorders
Keywords: Musculoskeletal disorders; shoulder rehabilitation; virtual reality
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with shoulder musculoskeletal disorders (Experimental): The study will involve 50 adults with shoulder musculoskeletal disorders. Eligible participants are those over 18 with significant shoulder pathologies, excluding individuals with neurological conditions, infections, inflammatory diseases, major previous shoulder surgeries, or pregnancy. After obtaining informed consent, baseline demographic and anthropometric data will be collected. Patients will be assessed by a clinician across four rehabilitation phases: T1 (0-4/6 weeks), T2 (6-12 weeks), T3 (12-20 weeks), and T4 (beyond 20 weeks). Each phase includes a shoulder examination followed by a 30-minute VR-based rehabilitation session, customized to the patient's physical characteristics.
  Interventions: Diagnostic Test: Shoulder Physical Examination; Procedure: Shoulder Rehabilitation in a Virtual Environment; Other: Usability assessment and presence and co-presence evaluation

INTERVENTIONS:
Diagnostic Test: Shoulder Physical Examination — shoulder physical examination is conducted to assess the patient's musculoskeletal condition and to track progress throughout the rehabilitation phases
Procedure: Shoulder Rehabilitation in a Virtual Environment — The rehabilitation protocol for shoulder disorders is executed using a Virtual Reality (VR) system, where patients perform customized exercises tailored to their physical characteristics.
Other: Usability assessment and presence and co-presence evaluation — The usability of the VR system, along with the sense of presence and co-presence during rehabilitation, is assessed using validated scales

SUMMARY:
Goal: The clinical investigation involves the evaluation of the usability level of the VR system, sense of presence, and co-presence during the execution of various rehabilitation exercises through specific questionnaires.

Participant Population: The study will enroll 50 patients with shoulder musculoskeletal disorders will be enrolled

Main Questions:

* How does the integration of Virtual Reality (VR) in rehabilitation programs impact the usability of the system for patients with shoulder musculoskeletal disorders?
* To what extent does the sense of presence experienced by patients using VR systems influence their motivation and adherence to rehabilitation exercises?
* How do patients with shoulder musculoskeletal disorders perceive the co-presence in VR rehabilitation scenarios, and how does it affect their overall treatment experience?

Participant Tasks:

* Shoulder Physical Examination
* Instructions to the patient on exercises to be performed using Oculus and selection of customizable settings on the VR app
* Execution of the protocol developed for shoulder rehabilitation in a virtual environment
* Evaluation of the usability of the VR system, sense of presence, and co-presence through different validated scales

DETAILED DESCRIPTION:
Musculoskeletal disorders are recognized globally as a primary cause of pain and physical disability. Among these, shoulder pathologies impose significant limitations, affecting patients' range of motion, quality of life, and daily functionality, often leading to substantial physical and occupational restrictions. Effective rehabilitation is essential for restoring functionality in patients with such disorders.

Traditionally, rehabilitative therapy relies on manual interventions by physiotherapists, which, while beneficial, can be hindered by logistical challenges, including limited accessibility to treatment facilities and professional availability. Additionally, at-home unsupervised exercises often suffer from low adherence due to reduced motivation and lack of engagement.

Technological advances in recent years have led to the development of novel rehabilitation strategies, particularly in virtual reality (VR) systems, which hold promising applications in musculoskeletal rehabilitation. VR provides a patient-centered, customizable approach that can adapt exercises to the individual's needs, making rehabilitation more engaging and accessible, especially for patients facing physical barriers to in-person care. Additionally, VR technology enables precise tracking of patient movements, offering an objective alternative to traditional assessments reliant on subjective observation and clinical scales.

Despite these advancements, the integration of VR into rehabilitative protocols for MSDs remains underexplored. This clinical study aims to assess the usability, sense of presence, and co-presence of VR systems in patients with shoulder musculoskeletal disorders across four rehabilitation phases. Evaluating these factors through validated questionnaires will provide critical insights into optimizing patient engagement and satisfaction, which are key to enhancing therapeutic outcomes and aligning rehabilitation interventions with patient-specific needs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shoulder musculoskeletal disorders
* Patients aged 18-75 years
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with insufficient cognitive and language functions to follow instructions provided by clinicians and/or experimenters involved in the project
* Patients who do exhibit impediments that could hinder the use of VR devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Usability Level of the VR System Using the System Usability Scale (SUS) | Across four rehabilitation phases: T1 (0-4/6 weeks), T2 (6-12 weeks), T3 (12-20 weeks), and T4 (beyond 20 weeks)
  The usability of the VR system during the execution of several rehabilitation exercises will be assessed using the System Usability Scale (SUS). The SUS is a widely used questionnaire that measures the overall usability of a system, based on a 10-item scale that assesses the ease of use, satisfaction, and functionality of the system from the user's perspective. Scores range from 0 to 100, with higher scores indicating better usability.

SECONDARY OUTCOMES:
Change in Sense of Presence Using the Igroup Presence Questionnaire (IPQ) | The sense of presence will be evaluated across four rehabilitation phases: T1 (0-4/6 weeks), T2 (6-12 weeks), T3 (12-20 weeks), and T4 (beyond 20 weeks)
  The sense of presence during the execution of rehabilitation exercises in the VR system will be assessed using the Igroup Presence Questionnaire (IPQ). The IPQ is a validated tool designed to measure the user's sense of immersion and involvement in a virtual environment. It includes multiple dimensions, such as spatial presence, engagement, and ecological validity, and provides insights into how "real" the virtual environment feels to the user.
Change in Co-Presence Using the Networked Minds Social Presence Inventory | The co-presence will be assessed across four rehabilitation phases: T1 (0-4/6 weeks), T2 (6-12 weeks), T3 (12-20 weeks), and T4 (beyond 20 weeks).
  Co-presence during the execution of rehabilitation exercises in the VR system will be assessed using the Networked Minds Social Presence Inventory. This inventory measures the user's perception of social interaction and the sense of being with others in a virtual environment. It evaluates factors such as interpersonal communication, social presence, and the degree to which users feel they share the virtual space with others.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The ownership of the data is of the promoter and shared with the investigators and will be managed according to the agreements between the participating institutions and with the researchers. Data Property belongs to Fondazione Policlinico Universitario Campus Bio-Medico. The personnel involved in this study will have access to all data. In agreement with the ICH-GCP, the principal investigator of the study agrees to produce a report on the study, share all the data collected as described in the Protocol, and ensure that the data are reported responsibly and consistently.
  The transmission or dissemination of data through scientific publications and/or presentations in congresses, conferences, seminars, and participation in multicenter studies will take place exclusively following a purely statistical processing of the same, or in any case, in an anonymous form.